CLINICAL TRIAL: NCT06647069
Title: A Phase 1, Open-label, Multiple Ascending Dose Basket Study to Evaluate the Safety and Activity of DR-0201 in Patients With Select Autoimmune Rheumatic Diseases
Brief Title: DR-0201 in Subjects With Autoimmune Diseases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dren Bio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DR-0201-AIM-001
Record Dates: First submitted 2024-10-16; First posted 2024-10-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: SLE; SLE (Systemic Lupus); CLE; Cutaneous Lupus; Sjogren's Syndrome; Primary Sjögren Syndrome; Dermatomyositis; Polymyositis; Scleroderma; SSc, Diffuse Sclerosis; dcSSc; Diffuse Cutaneous Systemic Sclerosis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Sjogren's Syndrome; Dermatomyositis; Polymyositis; Scleroderma, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- DL1 of DR-0201 (Experimental): Subjects in this arm will receive up to 6 months of dosing with dose level 1 of DR-0201
  Interventions: Drug: DR-0201
- DL2 of DR-0201 (Experimental): Subjects in this arm will receive up to 6 months of dosing with dose level 2 of DR-0201
  Interventions: Drug: DR-0201
- DL3 of DR-0201 (Experimental): Subjects in this arm will receive up to 6 months of dosing with dose level 3 of DR-0201
  Interventions: Drug: DR-0201
- DL4 of DR-0201 (Experimental): Subjects in this arm will receive up to 6 months of dosing with dose level 4 of DR-0201
  Interventions: Drug: DR-0201
- DL5 of DR-0201 (Experimental): Subjects in this arm will receive up to 6 months of dosing with dose level 5 of DR-0201
  Interventions: Drug: DR-0201
- DL6 of DR-0201 (Experimental): Subjects in this arm will receive up to 6 months of dosing with dose level 6 of DR-0201
  Interventions: Drug: DR-0201

INTERVENTIONS:
Drug: DR-0201 — DR-0201 is a bispecific antibody

SUMMARY:
This is a multi-center, open-label, multi-ascending dose study to evaluate the safety, tolerability, PK, PD, immunogenicity, and preliminary clinical response of DR-0201 following IV administration in subjects with SLE, CLE, pSS, PM/DM, and/or dcSSc.

ELIGIBILITY:
Inclusion Criteria:

1. American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) diagnosis of 1 of the following active autoimmune diseases: SLE or CLE (both must have CLASI > 8 at both screening and baseline visits); pSS; PM/DM (probable or definite); and/or dcSSc (of < 3 years duration).
2. Subjects with SLE, CLE, or dcSSc must be willing to undergo skin biopsies at baseline and 2 skin biopsies during the treatment period; subjects with pSS must be willing to undergo salivary gland biopsies at baseline and 2 salivary gland biopsies during the treatment period; subjects with PM must be willing to undergo muscle biopsies at baseline and 2 muscle biopsies during the treatment period; and subjects with DM must be willing to undergo muscle biopsies at baseline and 2 muscle biopsies during the treatment period or they may choose to undergo skin biopsies instead.
3. Between 18 and 75 years of age, inclusive, of either gender and of any race.
4. Stable, but active disease, such that in the opinion of the Investigator, it is unlikely that a change in the subject's therapeutic regimen would be required during the subsequent 3 to 4 months.
5. Photographs of skin lesions, when applicable, must be submitted for review to confirm that the lesions are suitable for punch biopsy and caused by SLE, CLE, or DM disease activity. Such confirmation by the Sponsor must be received prior to enrollment.
6. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF).
7. Use of a highly effective contraceptive measure (< 1% failure rate; see Section 13.1) for all non-sterilized males and all females of childbearing potential during study through 120 days after last DR-0201 dose. Females of childbearing potential need to have a negative serum pregnancy test within 7 days prior to the first dose of DR-0201. Females who are not of childbearing potential (i.e., who are considered to be post-menopausal [≥ 12 months of non-therapy amenorrhea] or surgically sterile [absence of ovaries and/or uterus]) are not required to have a pregnancy test or use contraception.

Exclusion Criteria:

1. Severe manifestation of the selected autoimmune rheumatic diseases under study that could impact participant safety, or is likely to require interventions that will affect investigational drug PD.
2. Receipt of super-high potency (e.g., clobetasol propionate) or high potency (e.g., fluocinonide) topical corticosteroids within 1 month prior to screening.
3. Received dose changes of mycophenolate mofetil, methotrexate, leflunomide, azathioprine, or nonsteroidal topical immunosuppressants within 28 days prior to Day 1 or dose changes of oral or topical corticosteroids within 14 days prior to Day 1.
4. Required regular use of medications known to cause, as a major side effect, dry mouth/eyes, and which have not been on a stable dose for at least 30 days prior to screening, or any anticipated change in the treatment regimen during the course of the study.
5. Receipt of any of the following medications within 6 months of Day 1: cyclophosphamide, leflunomide > 20 mg/day, abatacept.
6. Receipt of any mAb or experimental immunomodulator within 28 days or 5 published half-lives prior to Day 1, whichever is shorter.
7. Receipt of rituximab or other B cell depleting biologics within 6 months of Day 1.
8. Receipt of rituximab or other B cell depleting biologics without return of CD19 or CD20 count to above the LLN.
9. Receipt of alemtuzumab, bone marrow transplantation, stem cell transplantation, total lymphoid irradiation, chimeric antigen receptor T cell (CAR-T) or T cell vaccination therapy.
10. Known history of a primary immunodeficiency or an underlying condition such as known human immunodeficiency virus (HIV) infection, positive result for HIV infection, splenectomy, or any underlying condition that predisposes the subject to infection.
11. Subjects with AST > 2.5 × upper limit of normal (ULN), ALT > 2.5 × ULN, total bilirubin > 1.5 × ULN (unless due to Gilbert's syndrome), total immunoglobulin < 500 g/dL, neutrophil count < 1000/μL, platelet count < 85,000/μL, hemoglobin < 10 g/dL, glycosylated hemoglobin > 8%, total lymphocyte count < 300/μL, or glomerular filtration rate < 50 mL/min/1.73 m2.
12. History of a hypersensitivity reaction or anaphylaxis to a previous mAb or human immunoglobulin therapy.
13. Active infection or a history of serious infections as follows:

    1. Use of antimicrobials (antibacterials, antivirals, antifungals, or antiparasitic agents) for an infection within 30 days prior to the first dose of DR-0201. Topical treatments may be allowed at the Medical Monitor's discretion.
    2. History of opportunistic infections in the last 2 years.
    3. Recurrent or chronic infection, or other active infection, that in the opinion of the Investigator might cause this study to be detrimental to the subject.
    4. Symptomatic herpes zoster within 3 months prior to screening or recurrent herpes zoster or herpes simplex infections.
    5. History of tuberculosis (active or latent) irrespective of treatment status.
    6. Any history of viral hepatitis: hepatitis B virus, hepatitis C virus (HCV), hepatitis E virus. HCV is acceptable if HCV ribonucleic acid (RNA) is undetectable for at least 3 months after completion of direct-acting antiviral therapy.
14. Major surgery within 28 days prior to Day 1.
15. QT interval corrected for heart rate (QTc) > 480 msec, based on the mean of triplicate ECGs. The QTc is the QT interval corrected using Fridericia's formula (QTcF).
16. Evidence of significant, uncontrolled concurrent disease that could affect compliance with the study(e.g., chronic obstructive pulmonary disease).
17. Previous exposure to DR-0201.
18. Participation in a clinical trial and has received an investigational product within the following time period prior to screening in the current study: 3 months (for biologic therapies) or 1 month (for non-biologic therapies), 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is longer).
19. Unstable lifestyle factors (including but not limited to excessive alcohol use, heavy nicotine use, or substance abuse), to the extent that, in the opinion of the Investigator, they would interfere with the ability of a subject to complete the study.
20. Diagnosis or history of malignant disease within 5 years prior to baseline, with the exceptions of basal cell or squamous epithelial carcinomas of the skin that have been resected or cervical carcinoma in situ, with no evidence of recurrence within the 5 years prior to baseline.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events as assessed by CTCAE v5.0.(Safety and Tolerability) | Baseline to Day 239
  To determine the incidence and severity of adverse events as assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rothenberg, MD, PhD, Study Director — Dren Bio
Locations (10):
- Australia (2):
  - Dren Investigational Site, Coorparoo, Queensland
  - Dren Investigational Site, Melbourne, Victoria
- Bosnia and Herzegovina (2):
  - Dren Investigational Site, Mostar
  - Dren Investigational Site, Sarajevo
- Dren Investigational Site, Auckland, New Zealand
- South Africa (5):
  - Dren Investigational Site, Pretoria, Gauteng
  - Dren Investigational Site, Pretoria, Guateng
  - Dren Investigational Site, Polokwane
  - Dren Investigational Site, Pretoria
  - Dren Investigational Site, Vereeniging

IPD SHARING:
Plan to Share IPD: No